CLINICAL TRIAL: NCT06597214
Title: Intraoperative Warming: Comparison of Performance of the AVAcore Technologies warmUP™ Temperature Management System (WU-20) and the Arizant Bair Hugger Temperature Management System
Brief Title: Intraoperative Warming: Comparison of Two Temperature Management Systems
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Tampa General Hospital (Other)
Collaborators: TeamHealth (Unknown)
Responsible Party: Principal Investigator, Enrico, Emeritus Professor of Surgery, Tampa General Hospital
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: STUDY001814 Sleeve Blanket
Record Dates: First submitted 2024-09-06; First posted 2024-09-19 (Actual); Last update posted 2025-06-25 (Actual); Status verified 2025-06

CONDITIONS: Normothermia; Intraoperative Temperature; Anesthesia
Keywords: Forced-air warmers; perioperative temperature management

STUDY DESIGN:
Intervention Model Description: Prospective single-group assignment compared to a standard control.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- AVACore Technologies, Inc. warmUP Sleeve (Experimental): AVAcore Technologies's warmUP (WU-20) Temperature Management System was developed based on work with the Aquarius Medical Acrotherm device and prior human hypothermic subject data showing a rewarming rate of ~1ºC in 5 minutes when heat and vacuum application was tested. AVAcore Technologies received FDA acceptance of its Section 510(k) premarket notification for the warmUP (vH1) Temperature Management System in 2005. This product was used on over 100 patients in the US in 2005-2006 timeframe.
  Interventions: Device: AVACore Technologies, Inc. warmUP Sleeve; Device: Arizant Healthcare Bair Hugger®

INTERVENTIONS:
Device: AVACore Technologies, Inc. warmUP Sleeve — AVAcore Technologies's warmUP (WU-20) Temperature Management System was developed based on work with the Aquarius Medical Acrotherm device and prior human hypothermic subject data showing a rewarming rate of ~1ºC in 5 minutes when heat and vacuum application was tested. AVAcore Technologies received FDA acceptance of its Section 510(k) premarket notification for the warmUP (vH1) Temperature Management System in 2005. This product was used on over 100 patients in the US in 2005-2006 timeframe.
Device: Arizant Healthcare Bair Hugger® — The Arizant Healthcare Bair Hugger® Temperature Management System proposed for use in this study is a 'forced air' system providing convective warming via the circulation of warmed air through a specially designed blanket which is placed over a portion of the patient's body. This product has been in use in the US for over 20 years in a majority of hospitals.
  Other Names: Historical Control Group

SUMMARY:
The goal of this clinical trial is to compare two temperature management systems, the warmUP (WU-20) and the Bair Hugger®, in preventing perioperative hypothermia during surgeries. The study aims to determine whether the warmUP system is as effective as the Bair Hugger® in maintaining core body temperature.

The main questions this trial aims to answer are:

Does the warmUP system maintain intraoperative body temperatures as effectively as the Bair Hugger® during abdominal surgeries?

Does the warmUP system offer additional benefits, such as reduced bacterial dispersion compared to the Bair Hugger®?

Participants will:

Use either the warmUP or Bair Hugger® system during surgery Undergo abdominal surgeries lasting approximately 2.5 hours Have their core temperatures monitored to assess the effectiveness of the warming device

The study will evaluate whether the warmUP system provides equivalent temperature management with a smaller body surface area exposed, potentially offering advantages in surgical infection control.

DETAILED DESCRIPTION:
Mild perioperative hypothermia (core temperature 34-36ºC) occurs commonly during anesthesia and surgery as a result of a combination of factors: anesthetic induced impairment of thermoregulatory controls, internal redistribution of heat within the body, surgical site skin preparation and subsequent exposure to the 'cold' OR environment. Induction of general anesthesia causes marked changes in the distribution of body heat between the patient's core and periphery. An initial drop in core temperature of between 0.5 to 1.5ºC after induction is the result of internal core-to-periphery redistribution of body heat caused by a combination of anesthesia induced vasodilation and decreased thermoregulatory vasoconstriction. Continued thermal imbalance during anesthesia results from inability of metabolic heat production to overcome the heat loss.

The complications related to mild perioperative hypothermia have been documented in numerous studies and summarized in a 1999 article, "Maintaining intraoperative normothermia: a meta-analysis of outcomes with costs". Complications include reduced resistance to surgical wound infection, reduced platelet function, increased intraoperative loss of blood, increased incidence of ventricular tachycardia and morbid cardiac events, Additionally, the duration of postoperative recovery has also been shown to be prolonged by mild hypothermia.

Various warming methods, such as warm blankets, forced-air warmers and circulating water mattresses, are currently used to prevent and treat mild perioperative hypothermia. All are cutaneous approaches that rely on heating the peripheral tissues in order to increase the thermal core temperature. However, during certain surgical procedures such as laparatomy, a large section of the skin surface (ie., abdomen and part of the patient in contact with the OR table) is unavailable. This can limit the efficacy of methods such as forced-air warming which rely on a large skin surface for heat transfer. Thus, one criterion for an alternative non-invasive warming device is that the heat generated by that device reach its desired target; in the case of perioperative hypothermia, that target is the patient's thermal core.Grahn, et al determined that it would be feasible to combine subatmospheric pressure with a thermal load (heat) and then apply this combination to the body's own specialized heat transfer areas - the ArterioVenous Anastamoses (AVAs) -- found in the hands and the feet. By mechanically distending these specialized heat exchange vessels (the AVAs) through the application of negative pressure, heat can be transferred more efficiently to the body core.

AVAcore Technologies's warmUP (WU-20) Temperature Management System was developed based on work with the Aquarius Medical Acrotherm device (reference 510(k) number: K003368) and prior human hypothermic subject data showing a rewarming rate of ~1ºC in 5 minutes when heat and vacuum application was tested. AVAcore Technologies received FDA acceptance of its Section 510(k) premarket notification for the warmUP (vH1) Temperature Management System in 2005 (reference 510(k) number: K040911). This product was used on over 100 patients in the US in 2005-2006 timeframe.

The warmUP (WU-20) Temperature Management System proposed for use in this study is a minor modification to the vH1 System. The warmUP (WU-20) Temperature Management System is a released product covered with a Letter to File per an assessment based on FDA Guidance documents. The Arizant Healthcare Bair Hugger® Temperature Management System proposed for use in this study is a 'forced air' system providing convective warming via the circulation of warmed air through a specially designed blanket which is placed over a portion of the patient's body. This system has FDA acceptance (reference 510(k) number: K021473.) This product has been in use in the US for over 20 years in a majority of hospitals.

The primary objective is to determine if the AVAcore Technologies warmUP (WU-20) Temperature Management System is as effective as forcedair warming (Bair Hugger™, Arizant Healthcare, Eden Prairie, MN) for maintenance of intraoperative body temperature in patients undergoing abdominal surgery under general anesthesia. The critical endpoints to be evaluated in making this determination are 1) % of subjects with an average intraoperative esophageal temperature of ≥ 36º C and 2) % of subjects with an initial PACU sublingual temperature of ≥ 36º C.

Secondary objectives include 1) comparison of the core body temperatures

@ 60 minutes post anesthesia induction, 2) comparison of temperature trends during surgery and 3) comparison of the subjects' PACU temperature trends and hypothermic symptoms such as shivering.

ELIGIBILITY:
Inclusion Criteria:

* Subjects ages 18-80 who are having elective open abdominal surgery from 2-4 hours and requiring general anesthesia.

Exclusion Criteria:

* Patients who are not between ages 18-80
* Patients who are pregnant; all female patients of childbearing age will be given a pregnancy test on the day of surgery.
* Patients who have a break in skin integrity on extremity selected as application site
* Patients who have a history of allergic skin conditions
* Patients who have a history of bleeding disorders
* Patients who have a history of malignant hyperthermia

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2023-06-01 (Actual); Primary Completion 2025-05-15 (Actual); Study Completion 2025-05-15 (Actual)

PRIMARY OUTCOMES:
Initial Temperature | 60 minutes after induction of general anesthesia]
  Comparison of body temperature
Continuing Temperature trends | Recorded every 15 minutes from the start of administration of general anesthesia through end of administration of anesthesia; typically 4-5 hours.
  Comparison of body temperature throughout surgery
Post-operative temperature | 5 minutes after PACU admission
  Taking patient temperature whilst in recovery in the post-anesthesia care unit (PACU)

CONTACTS AND LOCATIONS:
Locations (1):
- Tampa General Hospital, Tampa, Florida, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Sessler DI. Mild perioperative hypothermia. N Engl J Med. 1997 Jun 12;336(24):1730-7. doi: 10.1056/NEJM199706123362407. No abstract available. PMID 9180091
- [Background] Davis AJ, Bissonnette B. Thermal regulation and mild intraoperative hypothermia. Curr Opin Anaesthesiol. 1999 Jun;12(3):303-9. doi: 10.1097/00001503-199906000-00008. PMID 17013328
- [Background] Sessler DI. Perioperative heat balance. Anesthesiology. 2000 Feb;92(2):578-96. doi: 10.1097/00000542-200002000-00042. PMID 10691247